CLINICAL TRIAL: NCT04528186
Title: The Effect of Healthy Eating Index on Maternal Thyroid Volume in Hyperemesis Gravidarum
Status: Completed | Type: Observational
Sponsor: Batman Training and Research Hospital (Other Government)
Collaborators: Baskent University (Other)
Responsible Party: Principal Investigator, Erhan Okuyan,M.D, Principal Investigator, Batman Training and Research Hospital
Other Study IDs: 289
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Healthy Diet; Thyroid Hypertrophy; Pregnancy Emesis
Keywords: Thyroid volume; , Healty eating index; , Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Low eating index scores(50-70)
  Interventions: Diagnostic Test: Maternal thyroid volume
- 2: High eating index scores(Above 70)
  Interventions: Diagnostic Test: Maternal thyroid volume

INTERVENTIONS:
Diagnostic Test: Maternal thyroid volume — Maternal thyroid volume measurement

SUMMARY:
The relationship between healthy eating index and maternal thyroid volume in patients with hyperemesis gravidarum is planned.

DETAILED DESCRIPTION:
In pregnant women(11-14 week) admitted to our hospital between the ages of 15-49; After the healthy eating index scores were made face to face by the dietician, it was planned to measure the maternal thyroid volume by the radiologist.Our hypothesis in our study is to determine whether healthy eating index has effects on thyroid volume and blood parameters.

ELIGIBILITY:
Inclusion Criteria:

* 15-49 years old pregnant women
* 11-14 Gestational week of pregnancy
* Do not use medication,
* have no history of illness,
* who participated in face-to-face meetings with a dietician,
* who want to be included in the study,
* No smoking or alcohol consumption
* Patients with a BMI between 15-25

Exclusion Criteria:

* Pregnant women who are not between 15-49 years old,
* patients with chronic disease such as heart disease, diabetes,
* Patients who do not agree to meet with a dietician, patients who do not agree to be included in the study,
* smoking and alcohol use --Morbid-obese patients (BMI greater than 25)

Ages: 15 Years to 49 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Pregnant women between the ages of 15-49 who apply to our hospital
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Impact on Maternal Thyroid volume measures | 11-14 gestational week of pregnancy,Healty eating index scoresLow than 60 vs Higher than 60)
  Maternal Thyroid volume measures

SECONDARY OUTCOMES:
Ketonuria, Notrophil / platelet ratio, TSH / ft3 ratio | 11-14 gestational week of pregnancy
  Comparision of low and High eating index groups(Under 60 (low),Above 60(High))

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Okuyan, Principal Investigator — Batman Maternity and Child Health Hospital
Locations (1):
- Batman Maternity and Child Health Hospital, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No